CLINICAL TRIAL: NCT05177926
Title: A Prospective, Multi-center, Cohort Study to Evaluate the Efficacy and Safety of Tenofovir Alafenamide (TAF) for Prevention of Mother-to-child Transmission of Hepatitis B Virus Among Pregnant Women With High Level HBV DNA
Brief Title: Preventing Mother-to-child Transmission of Hepatitis B Virus With Tenofovir Alafenamide (TAF)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Gilead Sciences (Industry); Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Principal Investigator, Jinlin Hou, Professor & Director, Nanfang Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Shield-TAF
Record Dates: First submitted 2019-12-31; First posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Hepatitis B, Chronic; Mother to Child Transmission
Keywords: hepatitis B virus; mother-to-child transmission; antiviral prophylaxis; Tenofovir Alafenamide
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Intervention Model Description: This is a single arm study, in which all participants will receive study drug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- antiviral prophylaxis with Tenofovir Alafenamide Fumarate (TAF) (Other): All participants will receive oral Tenofovir Alafenamide Fumarate 25mg, daily, at gestational 27-29 week until delivery.
  Interventions: Drug: antiviral prophylaxis with Tenofovir Alafenamide Fumarate

INTERVENTIONS:
Drug: antiviral prophylaxis with Tenofovir Alafenamide Fumarate — All participants will receive antiviral prophylaxis with Tenofovir Alafenamide Fumarate for preventing of Mother-to-child transmission of HBV

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Tenofovir alafenamide (TAF) for prevention of mother-to-child transmission of hepatitis B virus among pregnant women with high level HBV DNA.

DETAILED DESCRIPTION:
This is a single-arm multicenter, prospective, clinical study, aiming to evaluate the efficacy and safety of Tenofovir alafenamide (TAF) for prevention of mother-to-child transmission of hepatitis B virus among pregnant women with high level HBV DNA. 330 HBV-infected mothers with high level HBV DNA will be enrolled and receive Tenofovir alafenamide (TAF) for prevention of mother-to-child transmission of HBV. Demographic data, antiviral treatment history, pregnancy and labour history, co-morbidity, HBV serologic marker tests, HBV DNA tests, liver function tests, mode of delivery, neonatal characteristics (height, weight, head circumference, Apgar score and any major birth defect), breastfeeding and post vaccination serological test for infants at 7-12 months of age are collected. A mobile health application called "SHIELD" is used in this study to collect data and provide support for communication between mothers and their doctors. All laboratory test reports, questionnaires and other relevant information are uploaded into SHIELD.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman aged 20 to 35 years old
* 24-26 week of gestation
* HBsAg positive more than 6 months and HBeAg positive
* HBV DNA> 200,000 IU/ml
* Informed consent is signed voluntarily by both husband and wife
* Good compliance and able to be followed up as planned

Exclusion Criteria:

* Mothers co-infected with HCV and HIV
* Evidence of decompensated cirrhosis and liver cancer
* Mothers had other organ lesions which would affect patient compliance and follow-up plan
* Mothers had history of spontaneous abortion or their children had birth defect or congenital malformation
* Mothers received antiviral therapy within 6 months
* Mothers had history of kidney injury, CCr <50ml/min and urine protein test positive (>300mg/L)
* Mothers had history of other chronic diseases and had to take immunomodulators, cytotoxic drugs or hormonal drugs during pregnancy
* The infants' biological fathers are infected with HBV
* Symptoms of threatened abortion during early pregnancy
* ALT > 1×upper limit of normal (ULN), or TBIL ≥ 1×ULN or glomerular filtration rate (GFR) < 90 ml/min, or Albumin (ALB) < 25 g/L
* Fetal malformations detected by B-ultrasound during pregnancy
* Participating in other studies

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant woman is eligible for mother-to-child transmission study.
Enrollment: 330 (Estimated)
Dates: Start 2021-04-04 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of mother-to-child transmission of HBV | from enrollment to the last infant completes post vaccination serological test (PVST), assessed up to 32 months
  the number of HBV-infected infants relative to all participants enrolled or to all participants who complete follow-up

SECONDARY OUTCOMES:
Rate of birth defect of infants | from enrollment to the last mother delivery, assessed up to 24 months
  the number of infants with birth defect relative to all participants enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Jinlin Hou, Study Chair — Nanfang Hospital, Southern Medical University
Locations (13):
- China (13):
  - The First Affiliated Hospital of Jilin University, Changchun
  - The First People's Hospital of Foshan, Foshan
  - Guangdong Maternal and Child Care Hospital, Guangzhou
  - Guangzhou No. 8 People's Hospital, Guangzhou
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - The Fifth Affiliated Hospital of Southern Medical University, Guangzhou
  - Zhujiang Hospital, Southern Medical University, Guangzhou
  - Affiliated Hangzhou First People's Hospital, Zhejiang University School of Medicine, Hangzhou
  - Xixi Hospital of Hangzhou, Hangzhou
  - The Affiliated Nanjing Hospital of Nanjing University of Chinese Medicine (The Second Hospital of Nanjing), Nanjing
  - Shanghai Public Health Clinical Center, Shanghai
  - Shenzhen Baoan Maternal and Child Care Hospital, Shenzhen
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an

IPD SHARING:
Plan to Share IPD: No